CLINICAL TRIAL: NCT06624137
Title: Computationally, Electrophysiologically, and Qualitatively Characterizing Serotonergic Psychedelics; Transdiagnostic Therapeutic and Pro-Psychotic Effects
Brief Title: Computer Game, Qualitative, and MEG/EEG Assessment of Serotonergic Psychedelics
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Burroughs Wellcome (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000025076
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: OCD; Major Depressive Disorder (MDD); Alcohol Use Disorder (AUD); Healthy Volunteer; Migraine; PTSD; PTSD - Post Traumatic Stress Disorder; Addiction; Tobacco Use Disorder; Obsessive Compulsive Disorder (OCD); Opioid Use Disorder
Keywords: Psilocybin; DMT; N,N-dimethyltryptamine; Ayahuasca; Lysergic acid diethylamide; LSD; 5-MeO-DMT; O-methyl-bufotenin; eeg; meg; 5-Methoxy-N,N-Dimethyltryptamine
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism; Migraine Disorders; Stress Disorders, Post-Traumatic; Combat Disorders; Behavior, Addictive; Tobacco Use Disorder; Obsessive-Compulsive Disorder; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serotonergic Psychedelic Arm: Group (healthy or with psychological or neurological disorder) administered serotonergic psychedelic (psilocybin, DMT, LSD, 5-MeO-DMT, Ayahuasca, etc.) regardless of administration route.
  Interventions: Drug: Serotonergic Psychedelic
- Placebo Arm: Group (healthy or with psychological or neurological disorder) administered placebo (diphenydramine, saline, niacin, etc.) regardless of administration route.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serotonergic Psychedelic — Any serotonergic or "classic" psychedelic that exhibits mainly Serotonin 2A receptor (5-HT2AR) agonism and is judged to produce subjectively similar effects.
  Groups: Serotonergic Psychedelic Arm
Drug: Placebo — Matched Placebo
  Groups: Placebo Arm

SUMMARY:
The goal of this observational study is to learn how the brain's information processing changes during and following administration of serotonergic psychedelics (psilocybin, N,N-Dimethyltryptamine/DMT, Lystergic Acid Diethylamide/LSD, etc.) for people with and without mental illness receiving serotonergic psychedelics through any clinical trial at Yale University. The main questions it aims to answer are:

1. Do serotonergic psychedelics cause the brain to rely on new information more than previously learned information while under the influence? What about 1 day, 5-14 days, and 4-6 weeks after use?
2. Do serotonergic psychedelics cause long-lasting side-effects in how people perceive (see, hear, feel, etc.) the world and how easily people change their beliefs?
3. How does the brain's electrical activity change after using serotonergic psychedelics? How does the balance between excitation and inhibition change while under their effect?
4. Can changes in how the brain uses information predict who will benefit from a psychedelic and who will have side effects from psychedelics?

Researchers will compare with people given placebos to see what changes in brain processing are unique to serotonergic psychedelics.

Participants will have the opportunity to do some combination of the following:

1. Online computer assessments consisting of games and questionnaires that probe how participants think.
2. Magnetoencephalography (MEG) or electroencephalography (EEG) with eyes closed and with repeated clicks, images, or sensations delivered.
3. A magnetic resonance imaging (MRI) scan.
4. Semi-structured qualitative interviews about their experience after taking a serotonergic psychedelic recorded via Zoom.

DETAILED DESCRIPTION:
Mounting evidence suggests that serotonergic psychedelics (SPs; eg. psilocybin, LSD) reduce symptoms across many mental illnesses with rapid, sustained effects from single interventions. They also cause persisting, positive effects in the general population and those without mental illness. This improved wellness comes at the cost of acute psychosis-like effects, that sometimes persist in weakened forms or, rarely, as prolonged episodes of psychosis. Understanding the mechanism underlying these dual effects may help maximize therapeutic effect and minimize unwanted outcomes.

The reason SPs cause therapeutic change and also cause psychotic-like effects regardless of whether one has a mental illness may be because they alter the basic machinery that the brain uses to process all information. SPs seem to shift processing-in both how we perceive (seeing, hearing, etc.) and learn-to rely more on new, incoming information over previously learned information. Essentially, SPs shift the brain into an extreme learning mode that allows it to modify harmful thought patterns associated with many mental illnesses, but that may also be similar to the brain states of early psychosis.

Participants in this study will opt-in to complete various measures to be completed before, during, and after being administered a serotonergic psychedelic through a clinical trial at Yale University.

How participant's brains process information will be assessed by:

1. Playing 3-4 computer games that measure how people see, hear, and learn. These will be completed 1-30 days before receiving the serotonergic psychedelic, the day they receive the serotonergic psychedelic (once psychologically acceptable and permitted by relevant trial researchers), the day after, 5-14 days after, and 4-6 weeks after.
2. MEG or EEG to measure the brain activity responsible for representing new vs. old information-and structural MRI to determine where the activity is coming from. The MEG/EEG will be done the day before, day of, and day after administration of the serotonergic psychedelic. The MRI can be done before, after, or during the trial.

They behaviors that accompany these changes will be assessed by:

1. Validated, online questionnaires at the same time points as the computer games.
2. Semi-structured interviews about what participants' day-to-day experiences are like and how they have changed after taking a serotonergic psychedelic. These may be done 2-5 days after using a psychedelic, or at the same time that clinical trial staff do their interviews.

Participants participating in a trial with single-arm placebo-controlled study design that includes a placebo arm may only complete these measures around a placebo administration. Those in a trial with a crossover design may complete these measures twice (except for day 1-30 and 4-6 week time points). Those opting to complete open-label administrations after study completion may complete relevant time points.

The primary objectives are to:

1. Investigate how serotonergic psychedelics change brain reliance on new vs. old information in perception and belief-updating while under the influence.
2. Investigate how serotonergic psychedelic change brain reliance on new vs. old information in perception and belief updating at short and long-term follow-up.
3. Investigate whether serotonergic psychedelics cause side effects in people's perception, attention, and belief updating that are both healthy and psychosis-like.
4. Investigate how serotonergic psychedelics acutely alter excitation/inhibition (E/I) balance in the brain.
5. Investigate whether there are any persisting changes in resting state EEG power or E/I balance.

The secondary objectives are to:

1. Investigate whether changes in brain information processing can explain therapeutic effects of serotonergic psychedelics.
2. Investigate whether changes in brain information processing can predict who will respond positively to serotonergic psychedelics.
3. Investigate whether changes in brain information processing can explain psychotic-like side effects of serotonergic psychedelics.
4. Investigate whether changes in brain information processing can predict who will have stronger psychotic-like side effects from serotonergic psychedelics.
5. Investigate whether acute or persisting changes in E/I balance predict therapeutic or psychotic effects of serotonergic psychedelics.

ELIGIBILITY:
Inclusion Criteria:

* Participation in approved clinical protocol at Yale University involving potential administration of serotonergic psychedelics
* Absence of pre-existing psychotic symptoms

Exclusion Criteria:

* Current intoxication based on self-report
* Any neurological, medical or developmental problem that is known to impair cognition significantly based on self-report
* History of seizures based on self-report
* Contraindications for MR scanning including metallic implants of any kind, pacemakers and history of accidents with metal, claustrophobia (specific to those who will participate in MRI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 individuals who have consented to be administered serotonergic psychedelics through a clinical trial at Yale University.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Hierarchial Gaussian Filter (HGF)-estimated average precision-weighted prediction error change in the conditioned hallucinations and probabilistic reversal learning tasks | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants' trial-by-trial responses on auditory and visual conditioned hallucination (CH) tasks as well as a probabilistic reversal learning (PRL) task are fitted with an enhanced Hierarchial Gaussian Filter (eHGF) model of hierarchial belief updating under perceptual/informational uncertainty using eHGF package in Julia. Precision weighted prediction errors used to update the 2nd and 3rd levels are estimated for each trial for each individual. Average precision weighted prediction errors across all trials as well as trials with greatest changes (0 stimulus trials for CH tasks and the first 5 trials after reversal in PRL) will be calculated. Change relative to baseline will be calculated. Greater precision weighted prediction errors reflect a greater weighting of new compared to previously learned information and greater belief updating.
Auditory and visual conditioned hallucination rate change | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants indicate detection of an auditory tone or visual pattern within auditory or visual noise. These stimuli are paired with cross-modality cues, causing participants to subconsciously expect to detect the stimuli using pavlovian conditioning. This conditioning causes participants experience "conditioned hallucinations" where they perceive the stimuli when it is not present. Conditioned hallucination rate is calculated as number of trials in which no stimulus was present but participants indicated perceiving the stimulus divided by the total number of trials in which no stimulus was present.
  A greater conditioned hallucination rate indicates greater reliance on previously learned information over incoming sensory evidence and closely tracks state-level hallucination susceptibility.
Perseverative and jumping-to-conclusion error total change in probabilistic reversal learning task | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants choose one of three images over multiple trials and receive reward feedback (low vs. high) in the PRL task. Each image has different reward probabilities that are unknown to participants. Through trial and error, participants learn which image is most rewarding and aim to maximize winnings. Over time, reward probabilities reverse without warning, requiring participants to update their beliefs. Every trial is scored as a perseverative error, a jumping to conclusions error, or neither, and then total number of error types are counted. Perseverative error trials occur when participants select a high reward probability image after its reward probability switches and they receive negative feedback. Jumping to conclusions (JTC) errors occur when participants switch from the highest reward stimulus to a different stimulus when there has been no reversal.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) score change | 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16-item self-report questionnaire that captures life satisfaction over the past week. Each question is scored on a 5-point scale from 1 (Very Poor) to 5 (Very Good) that indicates the degree of enjoyment or satisfaction achieved during the past week relative to the particular activity or feeling described in the item. Scores range from 16 to 80. Higher score indicates higher quality of life.
Southampton Mindfulness Questionnaire (SMQ) score change | 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  The Southampton Mindfulness Questionnaire (SMQ) consists of 16 items, each scored on a seven-point Likert scale from 0 = "Strongly Disagree" to 6 = "Strongly Agree." It measures the degree to which individuals are able to bring mindfulness to challenging or distressing thoughts and feelings. The total score is obtained by summing all items and ranges from 0 to 96. Higher scores indicate greater mindfulness in response to distressing situations.
HGF-estimated ratio of perceptual belief-to-sensory evidence weighting change | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  In the auditory and visual conditioned hallucinations tasks, the Julia eHGF model will estimate a single parameter value "Nu" for each individual that captures the individual's ratio of perceptual belief weighting compared to sensory evidence weighting in perceptual inference. Nu is estimated, like precision errors, by inverting the model from participant choices at each stimulus strength.
  Higher Nu values indicate participants are more likely to rely on learned pavlovian associations rather than sensory evidence and thus report perceiving the stimulus rather than not (IE experience a conditioned hallucination).
Aberrant Salience Inventory (ASI) score change | 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  The Aberrant Salience Inventory (ASI) consists of 29 items, each scored on a dichotomous scale: 0 = "No" and 1 = "Yes." It measures a variety of experiences related to aberrant salience, which refers to the inappropriate assignment of importance or significance to irrelevant, everyday, incoming stimuli/noise. The total score is calculated by summing all 29 items (0-29 range). Higher scores indicating higher levels of aberrant salience.
Change in the exponent of the 1/f power spectrum law from resting state EEG | Period of peak drug effect and 1 day after drug administration
  Excitation/Inhibition (E/I) balance will be approximated by calculating the exponent of the 1/f power spectrum law from participants' processed EEG power spectra using the Fitting Oscillations and One-Over-F (FOOOF) package in python. Lower exponents indicate a shift towards excitation in E/I balance - hypothesized to reflect bottom-up noise.
Change in resting state delta, alpha, theta, low gamma, medium gamma, and high gamma bands | Period of peak drug effect and 1 day after drug administration
  At least 10 minutes of resting state M/EEG with eyes closed will be recorded at each time point. For recording during acute drug administration, a 10 minute epoch of highest data quality around peak drug effect will be selected. After preprocessing to remove common artifacts and/or non-resting segments (eg. when participant opened eyes, moved around, or talked with study monitors), data will be filtered via fast fourier transformation (FFT) into canonical delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), low gamma (25 to 40 Hz), medium gamma (40 to 65 Hz), and high gamma (65 to 85 Hz) bands, and then average power (amplitude2) will be calculated. Change from baseline will be calculated for each participant in each band.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) score change | 5-14 days post drug administration and 4-6 weeks post drug administration
  The Patient Health Questionnaire-9 (PHQ-9) consists of 9 items, each scored on a four-point scale from 0 = "Not at all" to 3 = "Nearly every day." It measures the severity of depressive symptoms over the past two weeks. The total score is calculated by summing all 9 items, with higher scores indicating more severe depression. Scores range from 0 to 27 and are typically interpreted as follows: 0-4 = minimal depression, 5-9 = mild, 10-14 = moderate, 15-19 = moderately severe, and 20-27 = severe depression.
Change in learning rate difference between noisy and volatile learning conditions in a probabilistic learning game | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants complete a probabilistic learning game in which they estimate where objects will fall from an unseen spaceship, receiving trial-by-trial feedback on the actual location of the falling object. The location of the falling objects are sampled from a series of normal distributions that vary by mean and standard deviation such that changing means corresponds to high environmental volatility and high standard deviation correspond to high noise. Every trial produces a prediction error between the participant guess of where the object will fall and the actual position. Learning rate (LR) is calculated on each trial by dividing the subsequent change in participant estimate by the difference in estimate and actual object location (the prediction error). Average LR for each of 5 levels will be calculated. Higher average LRs reflect greater weighting of prediction errors and learning from new information under each level's condition.
Change in jumping to conclusion and perseverative errors in a feedback-free probabilistic learning game | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants must guess which of 3 ponds a colored fish was drawn from. They can see the proportion of each color of fish in each pond. Without warning, the pond that fish are drawn from are switched. Trials in which participants select the pond from which fish were previously drawn after a new pond is being sampled from are perseverative errors. Trials in which a participant mistakenly believes that a selection of a rare fish from the pond represents a shift to a new pond are marked as jumping-to-conclusion (JTC) errors. Total perseverative and JTC errors are calculated for each participant. More perseverative errors indicates difficulty updating beliefs and overreliance on prior compared to new information. More JTC errors indicate oversensitivity to new information compared to previously learned information as well as difficulty distinguishing probabilistic noise from environmental volatility.
Reward and punishment learning rate changes in probabilistic reversal learning task | Immediately post drug administration (when psychologically acceptable), 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  Participants' behavior in the PRL task will also be modeled using Rescorla-Wagner reinforcement learning as a function of weighted updates from predictions errors. A single learning rate parameter - the weighting of prediction errors - is estimated for each participant. The model will also be run calculating two learning rates for each participant - differing by whether the prediction error was positive vs. negative (positive vs. negative outcome). Higher learning rates reflect greater reliance on new as opposed to previously learned information.
Psychedelic Change Questionnaire (PCQ-26) score change | 1 day post drug administration, 5-14 days post drug administration, and 4-6 weeks post drug administration
  The Psychedelic Experience Questionnaire-26 (PCQ-26) consists of 26 items, each scored on a seven-point Likert scale from 1 = "Very much improved" to 7 = "Very much worse," with 4 = "No change." It assesses the impact of a psychedelic experience across multiple domains, including emotional, cognitive, and perceptual changes, as well as changes in well-being and personal growth. The total score is calculated by summing all 26 items, with lower scores reflecting more positive and enduring changes after a psychedelic experience. Three factors are also scored the same way. Lower Factor 1 scores indicate more positive perceptions/cognitions/emotions that are often experience during the acute experience. Higher factor 2 scores indicate better physical states/functioning (eg. sleep, appetite, and sexuality). Higher factor 3 scores reflect prosocial emotions and motivations.

CONTACTS AND LOCATIONS:
Overall Officials: Maximillian S Greenwald, BA, Study Director — Yale University; Albert R Powers, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, Hamden, Connecticut
  - West Haven VA Medical Center, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to share individual participant data.